CLINICAL TRIAL: NCT07334080
Title: A Phase I, Open-Label, Randomized, Single-Dose, Crossover Study to Evaluate Food Effect and Relative Bioavailability of ECC4703 Formulations (F0, F1, F2, and F3) in Healthy Adults
Brief Title: ECC4703 Food Effect and Relative Bioavailability Study in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC0008
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Dysfunction-Associated Steatohepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ECC4703 F1 formulation (Experimental): Participants will receive a single dose of ECC4703 F1 high-fat or fasted state, followed by ECC4703 F1 fasted or high-fat state, respectively, in subsequent treatment periods
  Interventions: Drug: ECC4703 F1 formulation
- ECC4703 F2 formulation (Experimental): Participants will receive a single dose of ECC4703 F2 high-fat or fasted state, followed by ECC4703 F2 fasted or high-fat state, respectively, in subsequent treatment periods
  Interventions: Drug: ECC4703 F2 formulation
- ECC4703 F3 formulation (Experimental): Participants will receive a single dose of ECC4703 F3 high-fat or fasted state, followed by ECC4703 F3 fasted or high-fat state, respectively, in subsequent treatment periods
  Interventions: Drug: ECC4703 F3 formulation
- ECC4703 F0 formulation (Experimental): Participants will receive a single dose of ECC4703 F0 fasted state, followed by ECC4703 F1, F2 or F3 fasted in subsequent treatment periods
  Interventions: Drug: ECC4703 F0 formulation; Drug: ECC4703 F1 formulation; Drug: ECC4703 F2 formulation; Drug: ECC4703 F3 formulation

INTERVENTIONS:
Drug: ECC4703 F0 formulation — A single dose of ECC4703 F0
  Arms: ECC4703 F0 formulation
Drug: ECC4703 F1 formulation — A single dose of ECC4703 F1
  Arms: ECC4703 F0 formulation; ECC4703 F1 formulation
Drug: ECC4703 F2 formulation — A single dose of ECC4703 F2
  Arms: ECC4703 F0 formulation; ECC4703 F2 formulation
Drug: ECC4703 F3 formulation — A single dose of ECC4703 F3
  Arms: ECC4703 F0 formulation; ECC4703 F3 formulation

SUMMARY:
This is a Phase I, open-label, randomized, single-dose, 2-part study designed to evaluate the food effect and relative bioavailability of ECC4703 in healthy adult participants.

DETAILED DESCRIPTION:
Part 1 will include 3 cohorts of 16 participants each, completing 2 single-dose crossover periods to assess food effect on ECC4703 formulations (F1, F2, and F3). Part 2 of the study will enroll approximately 24 participants to compare selected formulations from Part 1 to formulation (F0), using an adaptive design to finalize sequence, treatment periods, and food conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants
* Age of 18 to 65 years
* BMI of 18.0 to 32.0 kg/m2 with a minimum body weight of 50.0 kg (110 lb) for males and 45.0 kg (99 lb) for females.
* Female participants of childbearing potential must have negative serum pregnancy test at screening and a negative serum or urine pregnancy test prior to the first dose of study drug; use at least 1 highly effective method of contraception (e.g., hormonal contraception, intrauterine device, bilateral tubal occlusion, or vasectomized partner with confirmed success) during the study and for at least 90 days after the last dose of study drug; and refrain from egg donation or fertility treatments during the same period.
* Female participants who are postmenopausal, confirmed by FSH test, or surgically sterile, confirmed by medical documentation, or agree to practice true abstinence
* Male participants agree to use contraception, or agree to practice true abstinence
* Not taking any medication within 14 days (or at least 5 half-lives whichever is longer) prior to Day 1 dosing, with the exception of stable-dose contraception, stable-dose hormonal replacement therapy, paracetamol at up to 2 g/day; or other medication, which in the opinion of the investigator and sponsor will not interfere with study assessments.
* No clinically significant findings in physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, clinical laboratory evaluations, concomitant medications, or medical/psychiatric history
* Able to understand and sign and date informed consent

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant, or breastfeeding during the study or within 90 days after the study.
* Concomitant participation in any investigational study of any nature
* Blood loss of ≥470 mL for non-physiological reasons (i.e., trauma, blood collection, blood donation) within 3 months prior to the first dose of study drug, plasma donation within 2 weeks prior to the first dose, platelet donation within 6 weeks prior to the first dose, or plans to donate blood during this study or within 1 month after the last dose of study drug.
* Clinically relevant acute or chronic medical conditions or diseases of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, immune or dermatologic systems
* Significant allergic reaction to active ingredients or excipients of the study drug
* Regularly uses tobacco or nicotine products, including e-cigarettes (>5 times per week) or has stopped using regular tobacco or nicotine products within the past 2 months.
* Unwilling to abstain from alcohol-containing products and/or xanthine/caffeine-containing products, including any food and beverages, within 48 hours prior to admission to the CRU on Day -1.
* Unwilling to abstain from grapefruit, grapefruit juice, and Seville oranges from 7 days prior to check-in on Day -1 until after their final follow-up visit.
* Unable to refrain from the use of any over-the-counter medications, prescription medications, nutritional supplements, or herbal medicines during the study, except for stable-dose contraception, stable-dose hormonal replacement therapy, paracetamol at up to 2 g/day; or other medication, which in the opinion of the investigator and sponsor will not interfere with study assessments.
* Any clinically significant abnormal findings in the participant's physical examination, laboratory tests, pregnancy test, urine drug screen, alcohol test, or medical history which in the opinion of the Investigator would prevent the participants from participating in the study.
* Has had clinically significant interventional therapies and/or hospitalization (surgery, paracentesis, etc.) within 6 months prior to the study, or plans to have any surgeries during the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
ECC4703 pharmacokinetic (PK) parameters AUC0-tlast | Up to Day 13
  Area under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non-Zero Concentration
ECC4703 PK parameters AUC0-inf | Up to Day 13
  Area under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
ECC4703 PK parameters Cmax | Up to Day 13
  Maximum observed plasma concentration
ECC4703 PK parameters tmax | Up to Day 13
  Time of the maximum observed plasma concentration
ECC4703 PK parameters AUC0-t | Up to Day 13
  Area under the plasma concentration-time curve up to the last measurable concentration
ECC4703 PK parameters AUC0-24 | Up to Day 13
  Area under the plasma concentration-time curve from time 0 to 24 hours post-dose
ECC4703 PK parameters AUCextr | Up to Day 13
  percentage of area under the concentration-time curve that is due to extrapolation from the last measurable concentration to infinity
ECC4703 PK parameters tlag | Up to Day 13
  lag time (time delay between dosing and first observed plasma concentration)
ECC4703 PK parameters t1/2 | Up to Day 13
  elimination half-life
ECC4703 PK parameters CL/F | Up to Day 13
  apparent clearance

SECONDARY OUTCOMES:
Number of participants with adverse events, with abnormal laboratory test results, abnormal ECGs, abnormal vital signs, and abnormal physical examinations | Up to Day 18
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examination
ECC4703 PK parameters AUC0-t | Up to Day 13
  area under the plasma concentration-time curve up to the last measurable concentration
ECC4703 PK parameters AUC0-24 | Up to Day 13
  Area under the plasma concentration-time curve from time 0 to 24 hours post-dose
ECC4703 PK parameters AUCextr | Up to Day 13
  percentage of area under the concentration-time curve that is due to extrapolation from the last measurable concentration to infinity
ECC4703 PK parameters tlag | Up to Day 13
  lag time (time delay between dosing and first observed plasma concentration)
ECC4703 PK parameters t1/2 | Up to Day 13
  elimination half-life
ECC4703 PK parameters CL/F | Up to Day 13
  apparent clearance

CONTACTS AND LOCATIONS:
Overall Officials: Eccogene Clinical Trials, Study Director — Eccogene
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No